CLINICAL TRIAL: NCT02709720
Title: Phase II Clinical Trial With Metronomic Oral Vinorelbine and Tri-weekly Cisplatin as Induction Therapy and Subsequent Concomitantly With Radiotherapy (RT) in Patients With Lung Cancer (NSCLC) Locally Advanced Unresectable
Brief Title: Study of Vinorelbine and Cisplatin as Induction Therapy With Radiotherapy in Patients With Unresectable NSCLC
Acronym: NORA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Lung Cancer Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 15/02_NORA; 2015-003312-21 (EudraCT Number)
Record Dates: First submitted 2016-02-02; First posted 2016-03-16 (Estimated); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Cancer Lung Disease; NORA; GECP 15/02; Metronomic administration
MeSH Terms: conditions — Lung Neoplasms | interventions — Vinorelbine; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 Experimental group (Experimental): 2 cycles of metronomic Vinorelbine 50 mg + cisplatin, followed by 2 cycles of Vinorelbine 30 mg + cisplatin concomitant with radiotherapy
  Induction chemotherapy:
  * Cisplatin: 80 mg/m2 day 1 every 21 days, for 2 cycles.
  * Metronomic oral vinorelbine: 50mg/day, 3 days of each week for 2 cycles.
  Concomitant chemotherapy and radiotherapy:
  * Cisplatin: 80 mg/m2 day 1 every 21 days, for 2 cycles.
  * Metronomic oral vinorelbine: 30mg/day, 3 days of each week for 2 cycles. 1 cycle equals 21 days
  Radiotherapy treatment:
  Patients will receive concomitant thoracic radiation therapy, using a technique three-dimensional conformal radiation therapy, using an accelerator linear that operates with energy rays ≥ 6 MV. The total target RTT dose will be 66 Gy in 33 daily fractions of 2 Gy, which will be prescribed in accordance with the document of ICRU reference 50 of ICRU.
  Interventions: Drug: Vinorelbine; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Vinorelbine — Cycle 1 and 2 50 mg/day, (Monday, Wednesday and Friday)
  Other Names: Navelbine
Drug: Cisplatin — Cycle 1 and 2 day 1, 80 mg/m2
Drug: Vinorelbine — Cycle 3 and 4 30 mg/day, (Monday, Wednesday and Friday)
  Other Names: Navelbine
Drug: Cisplatin — Cycle 3 and 4 day 1, 80 mg/m2
Radiation: Radiotherapy — concomitant therapy during cycles 3 and 4. Total dose: 66Gy

SUMMARY:
Phase II clinical trial with metronomic oral vinorelbine and tri-weekly cisplatin as induction therapy and subsequent concomitantly with radiotherapy (RT) in patients with lung cancer (NSCLC) locally advanced unresectable

DETAILED DESCRIPTION:
Hypothesis: At present, administration of concomitant chemotherapy and radiation therapy is considered a treatment of choice for patients with unresectable stage III tumor selected clinically.

There is at present a systemic considered standard treatment in combination with radical radiotherapy. Nor is it established a dose of standard radiation therapy, but it is known that should never be less than 60Gy57.

Vinorelbine has shown a strong radio-sensitizer in-vitro37 effect. In the phase II study, The combination of oral vinorelbine with cisplatin as induction therapy and then concomitantly with radiotherapy (66Gy) has provided very encouraging efficacy results. Recently in the vortex scheme cisplatin study with oral vinorelbine concomitant maintained with radiation from the second cycle of chemotherapy was tested.

It is therefore a priority in this segment pathology seeking treatment regimens that improve the effectiveness and toxicity. Metronomic chemotherapy started with the idea of administering a cytostatic divided doses, for an extended period without interruption, can provide the advantage of exposing patients to significant dose chemotherapy without worsening the toxicity profile. All this makes it an attractive treatment strategy, and can also maintain radio sensitizing effect during concomitance.

ELIGIBILITY:
Inclusion criteria:

* Patients with histologically confirmed recent non small cell lung cancer unresectable stage IIIA and IIIB.
* Perform a baseline positron emission tomography (PET-CT) to rule out the presence of distant disease and confirm that it is a non-NSCLC radical surgical treatment candidate.
* The positive mediastinal lymph nodes by PET-CT must be confirmed histologically. Mediastinal involvement may be considered without histologically observe when there is a mass of lymph nodes where the margins are not distinguished.
* At least one measurable lesion on computerized tomography (CT).
* Performance status 0-1.
* Life expectancy> 12 weeks.
* Age ≥18 years and ≤ 75 years.
* Right renal function: creatinine ≤ 1.5 mg / dl or creatinine clearance> 60 ml / min.
* Right hematologic function: hemoglobin> 10 g / dl, neutrophils ≥ 1500 / mm3 and platelets ≥ 100,000 / mm3.
* Right hepatic function: bilirubin ≤ 1.5 times the upper limit of each center, transaminases ≤ 2.5 above the normal limit.
* Right lung function without bronchodilators: defined by a forced expiratory volume in 1 second (FEV1)> 50% of predicted normal volume and lung diffusing capacity for carbon monoxide (DLCO)> 40% of predicted normal.
* The proportion of normal lung exposed to> 20 Gy RT (V20) shall be ≤ 35%.This must be fulfilled before the start of treatment cycle 3.
* Signature of informed consent.

Exclusion Criteria:

* Weight loss> 10% in the 3 months prior to study entry.
* Intestinal problems that do not ensure proper absorption of oral vinorelbine.
* Pregnant or lactating women. Women of childbearing potential should have a negative pregnancy test, and both men and women under this condition should take contraceptive measures throughout the study.
* symptomatic sensory neuropathy> grade 1 toxicity criteria according to the CTCAE v4.
* Comorbidities uncontrolled.
* syndrome of the superior vena cava.
* pleural or pericardial effusion: are both considered as indicative of metastatic disease unless proven otherwise. Those who still remain cytologically negative for malignancy, are exudates also be excluded. It may include those with pleural effusion visible on chest radiography or too small to perform diagnostic puncture safely.
* Known hypersensitivity to drugs with similar study drug structure.
* Previous treatment with anticancer drugs, previous surgery or thoracic radiotherapy for lung cancer or for other reasons.
* History of other malignancy treated properly within 5 years except carcinoma in situ of the cervix or breast skin and basal cell carcinoma.
* Concomitant treatment with other antineoplastic drug or investigational.
* Patients at any psychological, family, sociological or geographical that may hinder compliance with the study protocol and monitoring program.
* history of neurological or psychiatric disorders that impede a properly understanding of the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — Hospital Puerta de Hierro; Bartomeu Massutí, MD, Principal Investigator — Hospital General Universitario de Alicante; Teresa Morán, MD, Principal Investigator — Germans Trias i Pujol Hospital; José Luis González Larriba, MD, Principal Investigator — Hospital San Carlos, Madrid; Manuel Dómine, MD, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz; José Miguel Sánchez, MD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Ramón de las Peñas, MD, Principal Investigator — Hospital Provincial de Castellón; María Guirado, MD, Principal Investigator — Hospital Gnral de Elche; Dolores Isla, MD, Principal Investigator — Hospital Lozano Blesa; Raquel Marsé, MD, Principal Investigator — Hospital Son Espases; Mª Angeles Sala, MD, Principal Investigator — Hospital de Basurto; Juan Coves, MD, Principal Investigator — Hospital Son Llátzer; Ana Laura Ortega, MD, Principal Investigator — Hospital de Jaén; David Vicente, MD, Principal Investigator — Hospital Universitario Virgen Macarena; Regina Gironés, MD, Principal Investigator — Hospital LLuís Alcanyís; Alfredo Paredes, MD, Principal Investigator — Hospital de Donostia; Margarita Majem, MD, Principal Investigator — Hospital Sant Pau i de la Santa Creu; Sergio Vázquez, MD, Principal Investigator — Hospital Lucus Agustí
Locations (18):
- Spain (18):
  - Hospital General Universitario de Elche, Elche, Alicante
  - ICO-Badalona, Badalona, Barcelona
  - Hospital Provincial de Castellón, Castellon, Castelló
  - H. Son Espases, Palma de Mallorca, Mallorca
  - Hospital Lluís Alcanyís, Xàtiva, Valencia
  - Hospital de Basurto, Bilbao, Vizcaya
  - H.G.U. Alicante, Alicante
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - H. de Donostia, Donostia / San Sebastian
  - Hospital de Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - H. de la Princesa, Madrid
  - H.U. Puerta de Hierro, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - H. Clínico San Carlos, Madrid
  - H. Son Llàtzer, Palma de Mallorca
  - Hospital Virgen de La Macrena, Seville
  - Hospital Clínico Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Provencio M, Majem M, Guirado M, Massuti B, de Las Penas R, Ortega AL, Domine M, Marse R, Sala MA, Paredes A, Moran T, Vazquez S, Coves J, Larriba JLG, Sanchez JM, Vicente D, Farre N, Fornos LF, Zapata I, Franco F, Serna-Blasco R, Romero A, Isla D. Phase II clinical trial with metronomic oral vinorelbine and tri-weekly cisplatin as induction therapy, subsequently concomitant with radiotherapy (RT) in patients with locally advanced, unresectable, non-small cell lung cancer (NSCLC). Analysis of survival and value of ctDNA for patient selection. Lung Cancer. 2021 Mar;153:25-34. doi: 10.1016/j.lungcan.2021.01.005. Epub 2021 Jan 10. PMID 33453470
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: 2 cycles of metronomic Vinorelbine 50 mg + cisplatin, followed by 2 cycles of Vinorelbine 30 mg + cisplatin concomitant with radiotherapy
  Vinorelbine: Cycle 1 and 2 50 mg/day, (Monday, Wednesday and Friday)
  Cisplatin: Cycle 1 and 2 day 1, 80 mg/m2
  Vinorelbine: Cycle 3 and 4 30 mg/day, (Monday, Wednesday and Friday)
  Cisplatin: Cycle 3 and 4 day 1, 80 mg/m2
  Radiotherapy: concomitant therapy during cycles 3 and 4. Total dose: 66Gy
Period: Overall Study
Arm/Group | Experimental Group
Started | 68
Completed | 65
Not Completed | 3
Not completed — Non-compliance with inclusion criteria | 1
Not completed — Protocol Violation | 1
Not completed — Not take study medication | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Group
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 62 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 65
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 65
Smoking status [Count of Participants; unit: Participants]
  Non smoker | 3
  Former smoker | 27
  Smoker | 35
Body mass index [Median (Full Range); unit: kg/m^2] | 26.6 [16.2 to 42.9]
Weight [Count of Participants; unit: Participants]
  Under weight | 2
  Normal weight | 21
  Overweight | 25
  Obesity | 17
ECOG [Count of Participants; unit: Participants] — ECOG Performance Status Scale: It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability
  GRADES:
  ECOG 0: Fully active. ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours ECOG 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours ECOG 4: Completely disabled ECOG 5: Dead
  Participants
    ECOG 0 | 34
    ECOG 1 | 31
Histology [Count of Participants; unit: Participants]
  Squamous cell carcinoma | 27
  Adenocarcinoma | 29
  Large cell carcinoma | 1
  Adenosquamous carcinoma | 4
  Others | 2
  Not registered | 2
Stage [Number; unit: participants] — Staging is a classification where cancer is located, if or where it has spread and whether it's affecting other parts of the body.
  There are 5 stages for NSCLC:
  Stage 0:tumor hasn't grown into nearby normal lung tissues Stage I:small tumor that hasn't spread to any lymph nodes Stage II:medium tumor that hasn't spread to the nearby lymph nodes or N1 Stage III: cancer spread to the lymph nodes but haven't spread to other distant parts of the body Stage IV: cancer has spread to more than 1 area in the other lung, the fluid surrounding the lung or the heart, or distant parts of the body
  participants
    IIIA | 27
    IIIB | 38
Stage T [Count of Participants; unit: Participants] — In the TNM system:
  Primary tumor (T)
  * TX means that there is no information about the tumor or it cannot be measured.
  * T0 means that there is no evidence of a tumor.
  * Tis refers to a tumor "in situ." This means that the tumor is only found in the cells where it started. It has not spread to any surrounding tissue.
  * T1-T4 describe the size and location of the tumor, on a scale of 1 to 4. A larger tumor or a tumor that has grown deeper into nearby tissue will get a higher number. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    TX | 1
    T1 | 5
    T2 | 10
    T3 | 13
    T4 | 36
Stage N [Count of Participants; unit: Participants] — Regional lymph nodes (N) NX: Cancer in nearby lymph nodes cannot be measured. N0: No regional lymph node metastases N1: Metastasis in ipsilateral peribronchial and/or ipsilateral hilar lymph nodes and intrapulmonary nodes, including involvement by direct extension N2: Metastasis in ipsilateral mediastinal and/or subcarinal lymph node(s) N3: Metastasis in contralateral mediastinal, contralateral hilar, ipsilateral or contralateral scalene, or supraclavicular lymph node(s)
  Participants
    N0 | 5
    N1 | 7
    N2 | 35
    N3 | 18
Stage M [Count of Participants; unit: Participants] — Distant metastasis (M)
  MX: Metastasis cannot be measured. M0: Cancer has not spread to other parts of the body. M1: Cancer has spread to other parts of the body.
  Participants
    M0 | 65
    M1 | 0
Electrocardiogram [Number; unit: participants]
  Not done | 2
  Normal | 54
  Not normal | 9
Respiratory functional tests [Number; unit: participants]
  Normal | 64
  Not normal | 1
Compliance [Number; unit: participants]
  Treatment completed | 51
  Treatment not completed | 14
Cycles [Count of Participants; unit: Participants]
  Cycle 1 to Cycle 4 completed | 51
  Cycle 1 to Cycle 3 completed | 2
  Cycle1 and Cycle 2 completed and C3 incompleted | 1
  Cycle 1 and Cycle 2 completed | 6
  C1 completed and C2 incompleted | 1
  Cycle 1 completed | 2
  Cycle 1 incompleted | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: To evaluate the efficacy in terms of progression-free survival (PFS) of oral metronomical vinorelbine and cisplatin as an induction treatment and then with concomitant radiotherapy. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions The PFS is defined as the time from the moment of patient inclusion to the documentation of progression or death from any cause (patients who die without evidence of progression, will be considered events on the date of death).
Time Frame: From patient inclusion up to the date of first documented progression or date of death from any cause, whichever came first, up to 24 months.
Population: All study patients will be included and analysed in the intention-to-treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Group
Number analyzed (Participants) | 65
months | 11.5 [9.6 to 15.4]

2. Secondary Outcome: Objective Response Rate 6 Month
Description: The objective response rate will be calculated from the sum of the number of patients whose best response is complete response, partial response and stable disease divided by the total number of patients eligible for the analysis. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: From the start of the treatment of the patient to 6 month afther the treatment end
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Group
Number analyzed (Participants) | 65
percentage of participants | 78.1 [64.6 to 86.9]

3. Secondary Outcome: Overall Survival (Estimated)
Description: Overall survival will be measured from the date of patient inclusion until death or loss of follow-up. In patients who have not died, the duration of survival will be censored on the date of the last contact if the patient causes loss of follow-up or on the date of the latest news.
Time Frame: From the date of randomization until end of follow up or death, up to 24 months.
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Experimental Group
Number analyzed (Participants) | 65
Month | 35.6 [24.4 to 46.8]

ADVERSE EVENTS:
Time Frame: 25 months
Arm/Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 2/65
Serious Adverse Events (participants affected / at risk) | 10/65
Other Adverse Events (participants affected / at risk) | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=65)
Visceral arterial ischemia (Vascular disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 (3)
Renal insufficiency (Renal and urinary disorders) | 4 (4)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=65)
Anemia (Blood and lymphatic system disorders) | 33 (33)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 22 (22)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 16 (16)
Esophagitis (Gastrointestinal disorders) | 23 (23)
Gastritis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 51 (51)
Fatigue (General disorders) | 26 (26)
Edema limbs (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Creatinine increased (Blood and lymphatic system disorders) | 3 (3)
Neutrophil count decreased (Blood and lymphatic system disorders) | 30 (30)
Platelet count decreased (Blood and lymphatic system disorders) | 12 (12)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 11 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hipocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hipomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT02709720/Prot_SAP_000.pdf